CLINICAL TRIAL: NCT00118105
Title: A Phase II Trial of Neoadjuvant Capecitabine, Oxaliplatin, and Bevacizumab for Resectable Colorectal Metastases in the Liver
Brief Title: S0408: Capecitabine, Oxaliplatin, and Bevacizumab in Pts Undergoing Surgery for Liver Mets From Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Budget Constraints
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000433491; S0408 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy + Surgery + Chemotherapy (Experimental): Preoperative Neoadjuvant Chemotherapy
  * Bevacizumab, 7.5 mg/kg, IV, Day 1 of cycles 1,2,3
  * Oxaliplatin, 130 mg/m^2, IV, Day 1 of cycles 1,2,3,4
  * Capecitabine, 1,700 mg/m^2/day divided, PO at 12 hr intervals, Days 1-14 of cycles 1,2,3,4
  Conventional surgery: After 4 cycles of chemotherapy
  Postoperative Neoadjuvant Chemotherapy
  * Bevacizumab, 7.5 mg/kg, IV, Day 1 of cycles 1,2,3,4
  * Oxaliplatin, 130 mg/m^2, IV, Day 1 of cycles 1,2,3,4
  * Capecitabine, 1,700 mg/m^2/day divided, PO at 12 hr intervals, Days 1-14 of cycles 1,2,3,4
  Interventions: Biological: bevacizumab; Drug: capecitabine; Drug: oxaliplatin; Procedure: conventional surgery

INTERVENTIONS:
Biological: bevacizumab — Preoperative: 7.5 mg/kg, IV, Day 1 of cycles 1,2,3 Postoperative: 7.5 mg/kg, IV, Day 1 of cycles 1,2,3,4
  Other Names: Avastin; NSC-704865
Drug: capecitabine — Pre & Post Operative: 1,700 mg/m^2/day, PO at 12 hr interval, Days 1-14 of cycles 1,2,3,4
  Other Names: Xeloda; NSC-712807
Drug: oxaliplatin — 130 mg/m^2, IV, Day 1 of cycles 1,2,3,4
  Other Names: NSC-266046
Procedure: conventional surgery — Resection

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving capecitabine and oxaliplatin together with bevacizumab before and after surgery may be an effective treatment for liver metastases.

PURPOSE: This phase II trial is studying how well giving capecitabine and oxaliplatin together with bevacizumab works in treating patients who are undergoing surgery for liver metastases due to colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the proportion of patients with resectable hepatic metastases secondary to colorectal cancer who undergo surgical resection and achieve a R0 resection after treatment with neoadjuvant capecitabine, oxaliplatin, and bevacizumab.
* Determine the probability of non-progression (i.e., stable disease or response [complete and partial, confirmed and unconfirmed]) in patients treated with this regimen.
* Compare the proportion of patients treated with this regimen who undergo surgical resection and those who achieve a R0 resection with that described in the literature.
* Determine overall survival and disease-free survival of patients treated with this regimen.
* Determine response by positron emission tomography in patients treated with this regimen.
* Correlate clinical outcome with expression of biomarkers (e.g., thymidylate synthase, dihydropyrimidine dehydrogenase, thymidine phosphorylase, excision repair cross complementing 1, and hTERT) and telomere length in patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Neoadjuvant therapy: Patients receive bevacizumab* IV over 30-90 minutes and oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

NOTE: *Bevacizumab is administered during courses 1-3 of neoadjuvant therapy.

* Surgery: Approximately 3-4 weeks after completion of neoadjuvant therapy, patients are evaluated. Patients with unresectable disease are removed from the study. Patients with resectable disease undergo surgical resection of liver metastases within 4-6 weeks after completion of neoadjuvant therapy.
* Adjuvant therapy: Beginning at least 28 days after surgical resection, patients with at least stable disease after completion of neoadjuvant therapy receive 4 courses of adjuvant bevacizumab**, oxaliplatin, and capecitabine as in neoadjuvant therapy.

NOTE: **Bevacizumab is administered during courses 1-4 of adjuvant therapy.

After completion of study treatment, patients are followed every 4 months until disease progression and then every 6 months for up to 3 years from study entry.

PROJECTED ACCRUAL: Approximately 35-65 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hepatic metastases secondary to colorectal cancer by percutaneous hepatic biopsy
* Resectable hepatic metastases by any of the following:

  * Minor resection (i.e., less than a hemihepatectomy)
  * Major resection (i.e., hemihepatectomy or extended hepatectomy)
  * Bilobar resection (including atypical resection)
* Synchronous primary tumor and hepatic metastases allowed
* Radiologic evidence of hepatic metastases by multiphasic contrast-enhanced spiral CT scan
* Resectable primary colorectal cancer that is in place allowed
* Measurable disease
* No evidence of extrahepatic metastases by chest x-ray or CT scan of the chest

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin ≥ 9.0 g/dL
* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3

Hepatic

* Bilirubin ≤ 2 times upper limit of normal (ULN)
* SGOT or SGPT ≤ 2.5 times ULN

Renal

* Creatinine clearance ≥ 60 mL/min
* Urine protein/creatinine ratio < 1 OR
* Urine protein < 1 g by 24-hour urine collection

Cardiovascular

* No uncontrolled hypertension (i.e., blood pressure > 150/90 mm Hg)

  * History of hypertension allowed provided it is well controlled on a stable regimen of anti-hypertensive therapy
* No arterial thromboembolic event within the past 12 months, including any of the following:

  * Transient ischemic attack
  * Cerebrovascular accident
  * Unstable angina
  * Myocardial infarction
* No peripheral vascular disease ≥ grade 2

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No pre-existing peripheral neuropathy ≥ grade 2
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 6 months since prior adjuvant chemotherapy for the primary tumor
* No prior systemic chemotherapy for metastatic disease
* No prior hepatic artery infusion chemotherapy for metastatic disease

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for metastatic disease

Surgery

* More than 7 days since prior colonoscopy or fine needle aspiration
* More than 28 days since prior major invasive surgery or open biopsy

Other

* At least 4 weeks since prior and no concurrent sorivudine or brivudine
* No prior radiofrequency ablation for metastatic disease
* No prior cryotherapy for metastatic disease
* No other prior ablative techniques for metastatic disease
* No concurrent cimetidine

  * Concurrent ranitidine or other drug from a different antiulcer class allowed
* No concurrent oral anticoagulation for treatment of thrombosis

  * Concurrent warfarin (1 mg) to maintain patency of central venous catheter allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with R0 resection after treatment | 16-18 weeks from registration
Probability of nonprogression (i.e., stable disease or response [complete and partial, confirmed and unconfirmed]) | 12 weeks from registration
Comparison of patients achieving R0 resection with literature | 16-18 weeks from registration
Overall survival | Up to 3 years
Disease-free survival | Up to 3 years
Positron emission tomography response | Registration and 12 weeks
Correlation of clinical outcome with expression of biomarkers and telomere length | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Nicolas Vauthey, MD, Principal Investigator — M.D. Anderson Cancer Center; Robert de W. Marsh, MD, Principal Investigator — University of Florida; Cathy Eng, MD, Principal Investigator — M.D. Anderson Cancer Center; Henry Q. Xiong, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center; Kevin G. Billingsley, MD, Principal Investigator — OHSU Knight Cancer Institute; Steven A. Curley, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (46):
- United States (46):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazooaa, Michigan
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Frontier Cancer Center, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Danville Regional Medical Center, Danville, Virginia
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Background] Abdalla EK, Eng C, Madary A, Vauthey JN; Southwest Oncology Group 0408. Southwest Oncology Group 0408: Phase II trial of neoadjuvant capecitabine/oxaliplatin/bevacizumab for resectable colorectal metastases in the liver. Clin Colorectal Cancer. 2006 Mar;5(6):436-9. doi: 10.3816/ccc.2006.n.015. No abstract available. PMID 16635283